CLINICAL TRIAL: NCT01484678
Title: Magnetic Resonance Imaging and Biomarkers for Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Oregon Health and Science University (Other); Children's Hospital of Philadelphia (Other); Shriners Hospitals for Children (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201700056-N; R01AR056973 (NIH); 176-2010 (Other: Univeristy of Florida); OCR16243 (Other: University of Florida)
Record Dates: First submitted 2011-10-10; First posted 2011-12-02 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Magnetic Resonance Spectroscopy; Magnetic Resonance Imaging; Muscle
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Saliva samples collected, and a one time Muscle Biopsy in Becker MD subjects and matched controls only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age Matched Controls: Age matched non-affected (non-DMD) boys * This arm is full
  Age matched non-affected men, matched for men with Becker MD *Recruiting
- Boys/Men with DMD: This group will include ambulatory and non-ambulatory boys/men with Duchenne Muscular Dystrophy ranging from 5-30 years old. *Recruiting
- Adults with Becker MD: This group will include ambulatory and non-ambulatory men with Becker Muscular Dystrophy ranging from 18-62 years old. * Recruiting

SUMMARY:
The purpose of this research study is to determine the potential of magnetic resonance imaging, spectroscopy, and whole body imaging to monitor disease progression and to serve as an objective outcome measure for clinical trials in Muscular Dystrophy (MD).

The investigators will compare the muscles of ambulatory or non-ambulatory boys/men with DMD with muscles of healthy individuals of the same age and monitor disease progression in those with DMD over a 5-10 year period. The amount of muscle damage and fat that the investigators measure will also be related to performance in daily activities, such as walking and the loss of muscle strength. In a small group of subjects the investigators will also assess the effect of corticosteroid drugs on the muscle measurements.

Additionally, the investigators will map the progression of Becker MD following adults with this rare disease. The primary objective is to conduct a multi-centered study to validate the potential of non-invasive magnetic resonance imaging and magnetic resonance spectroscopy to monitor disease progression and to serve as a noninvasive surrogate outcome measure for clinical trials in DMD and BMD. The secondary objective is to characterize the progressive involvement of the lower extremity, upper extremity, trunk/respiratory muscles in boys/men with DMD and BMD guiding clinical trials.

DETAILED DESCRIPTION:
The overall objective of this proposal is to validate the potential of noninvasive magnetic resonance imaging (MRI) and spectroscopy (MRS) to monitor disease progression and to serve as an outcome measure for clinical trials in muscular dystrophies. Duchenne muscular dystrophy (DMD) is one of the most devastating genetically linked neuromuscular diseases and is characterized by the absence of dystrophin, resulting in progressive muscle weakness, loss of walking ability and premature death. Despite the poor prognosis therapeutic interventions have been lacking, and outcome measures for clinical trials have been limited to measures of muscle function, quality of life, serum biomarkers of muscle breakdown and invasive muscle biopsies. Closely related to DMD, Becker muscular dystrophy (BMD) has also been largely neglected in therapeutic development, due to its heterogeneity, small patient population, lack of outcome measures and uncertainty surrounding the patterns of disease progression, which may be mutation-dependent. Additional quantitative outcome measures that are noninvasive and sensitive to changes in muscle structure and composition are needed to facilitate the rapid translation of promising new interventions from preclinical studies to clinical trials in both forms of muscular dystrophy. As such, this project targets the development and validation of magnetic resonance as a noninvasive biomarker of disease progression in muscular dystrophy. Using a multi-site research design this study will characterize the intramuscular lipid content, cellular muscle damage and contractile area in the lower and/or upper extremity muscles of 200 ambulatory or non-ambulatory boys/men with DMD, 105 ambulatory or non-ambulatory men with BMD, and 110 healthy age matched boys/men using a combination of sophisticated MRI and MRS technologies. The trunk and respiratory muscles will be characterized in a subgroup of subjects (80 DMD, 20 BMD and 10 controls). In order to assess the sensitivity of each MR measure individually as well as composite MR measures (combination of muscles) to disease progression, all boys/men with DMD or BMD will be re-evaluated in yearly or 6 month intervals. The predictive outcome value of MRI/MRS will be further evaluated by determining the relationship between changes in MR measures and loss in muscle strength and/or functional ability. Using MRI/MRS we will also examine the effect of initiating corticosteroid treatment on skeletal muscle characteristics and composition. Examination of muscles in BMD patients will allow us to increase our understanding of how much dystrophin is needed to protect the muscle. To this end we will specifically examine the relationship between the MR phenotype (e.g. fast or slow increases in fat fraction) and dystrophin mutations, dystrophin expression and other histological markers. Finally, to ensure the rigor of this study we will examine the day-day reproducibility, inter MR system reproducibility and inter-validate the MR measures using localized MRS (golden standard). We anticipate that the MR techniques developed and validated in this study will be suitable for clinical trials in a wide range of muscular dystrophies and other neuromuscular diseases. In addition, MR characterization may serve as a powerful tool to further advance our understanding of the pathogenesis of muscular dystrophy and help guide the design of future trials.

ELIGIBILITY:
Inclusion Criteria for boys with DMD:

1. Ambulatory and non-ambulatory males (ages 5-30 at baseline testing) previously diagnosed with DMD based on:

* clinical features with onset of symptoms before age five
* elevated serum creatine kinase level or
* absence of dystrophin expression, as determined by immunostain or western blot (<2%) and/or DNA confirmation of a dystrophin mutation *Subjects will not be excluded based on corticosteroid treatment or other clinical trials

Inclusion Criteria for adults with Becker MD:

1. Ambulatory males (ages 18-62) without disease or injury to the lower extremities
2. Specific recruitment of a subset of individuals with deletion mutations in the dystrophin gene involving either exon 51 or exon 45.

Inclusion Criteria for age matched controls for Becker MD subjects:

1. Ambulatory males (ages 18-62) without disease or injury to the lower and/or upper extremities will be eligible to participate in this study

Exclusion Criteria:

1. Males with a contraindication to an MR examination
2. Males with unstable medical problems
3. Males who are not able to cooperate during testing
4. Males with a secondary condition that may impact muscle metabolism, muscle function or functional ability (i.e. cerebral palsy, endocrine disorders, mitochondrial disease)
5. Daytime ventilation
6. Implantable Cardioverter Defibrillator- (ICD) or pace maker
7. Healthy boys/men who participate in competitive sports specific training in excess of 8 hours per week

Ages: 5 Years to 62 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects are recruited from across the country. Investigators have a website (www.imagingNMD.org) and advertise the study nationally through list serves. The study will be advertised at the website of non-profit MD organizations. General information will be emailed to faculty and colleagues around the country. Fliers and brochures will be distributed in participating local clinics, MDA clinics, non-profit organizations, local neuromuscular clinics, and in strategic locations in associated hospitals. Age-matched healthy men will be recruited to match subjects with Becker MD from local and university communities. Individuals interested in this study are asked to contact the site clinical coordinator, who will complete a telephone screening interview to assess eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intramuscular lipid up to 3-10 years | Change in baseline up to 3-10 years
  In BMD and DMD, the from baseline in intramuscular lipid of upper/ lower extremity and trunk/respiratory muscles, as well as composite measures.
  MR measures of intramuscular lipid will be measured in yearly intervals for a period up to 3-10 years.
Change from baseline in muscle T2 up to 3 months in DMD | Change in baseline up to 3 months
  In a subgroup of subjects the effect of corticosteroids on muscle T2 will be measured at 3 and 6 months. Muscle T2 is a noninvasive marker of muscle damage/inflammation and will be measured using MR. This substudy requires its own Primary and Secondary Outcome measures.
Correlation between MR measures of intramuscular lipid, functional endpoints and histological markers. | Through study completion, an average of 1 year
  In both BMD and DMD, the correlation between MR measures and functional endpoints will be determined, as well as the ability of MR measures to predict future change and loss in function.

SECONDARY OUTCOMES:
Change from baseline in muscle T2 up to 5-10 years | Change in baseline up to 5-10 years
  Muscle T2 will be measured in the lower extremity and/or upper extremity muscles using MR at yearly intervals up to 5-10 years.
  We will report the change for each year interval.
Change from baseline in muscle contractile area up to 5-10 years | change in baseline up to 5-10 years
  Muscle contractile area will be measured in the lower extremity and/or upper extremity muscles using MR at yearly intervals up to 5 years. We will report the change for each year interval.
Change from baseline in muscle T2 at 6 months | Change in baseline up to 6 months
  In a subgroup of subjects the effect of corticosteroids on muscle T2 will be measured at 3 and 6 months. Muscle T2 is a noninvasive marker of muscle damage/inflammation and will be measured using MR. This substudy requires its own Primary and Secondary Outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: William Rooney, PhD, Principal Investigator — Oregan Health and Science University; H. Lee Sweeney, PhD, Principal Investigator — University of Florida; Krista Vandenborne, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Willis AB, Zelikovich AS, Sufit R, Ajroud-Driss S, Vandenborne K, Demonbreun AR, Batra A, Walter GA, McNally EM. Serum protein and imaging biomarkers after intermittent steroid treatment in muscular dystrophy. medRxiv [Preprint]. 2024 Jun 16:2024.06.14.24308858. doi: 10.1101/2024.06.14.24308858. PMID 38947030
- [Background] Muntoni F, Signorovitch J, Sajeev G, Done N, Yao Z, Goemans N, McDonald C, Mercuri E, Niks EH, Wong B, Vandenborne K, Straub V, de Groot IJM, Tian C, Manzur A, Dieye I, Lane H, Ward SJ, Servais L; PRO-DMD-01 study investigators; Association Francaise contre les Myopathies; UK NorthStar Clinical Network; ImagingDMD investigators; cTAP. Meaningful changes in motor function in Duchenne muscular dystrophy (DMD): A multi-center study. PLoS One. 2024 Jul 10;19(7):e0304984. doi: 10.1371/journal.pone.0304984. eCollection 2024. PMID 38985784
- [Background] Ikelaar NA, Barnard AM, Eng SWM, Hosseini Vajargah S, Ha KCH, Kan HE, Vandenborne K, Niks EH, Walter GA, Spitali P. Large scale serum proteomics identifies proteins associated with performance decline and clinical milestones in Duchenne muscular dystrophy. medRxiv [Preprint]. 2024 Aug 7:2024.08.05.24311516. doi: 10.1101/2024.08.05.24311516. PMID 39148831
- [Background] Kim J, Morales JF, Kang S, Klose M, Willcocks RJ, Daniels MJ, Belfiore-Oshan R, Walter GA, Rooney WD, Vandenborne K, Kim S. A model-informed clinical trial simulation tool with a graphical user interface for Duchenne muscular dystrophy. CPT Pharmacometrics Syst Pharmacol. 2025 Nov;14(11):1765-1774. doi: 10.1002/psp4.13246. Epub 2024 Oct 3. PMID 39360574
- [Background] Jenkins BM, Dixon LD, Kokesh KJ, Zingariello CD, Vandenborne K, Walter GA, Barnard AM. Skeletal muscle symptoms and quantitative MRI in females with dystrophinopathy. Muscle Nerve. 2024 Nov;70(5):988-999. doi: 10.1002/mus.28235. Epub 2024 Sep 2. PMID 39221574
- [Background] Akima H, Lott D, Senesac C, Deol J, Germain S, Arpan I, Bendixen R, Lee Sweeney H, Walter G, Vandenborne K. Relationships of thigh muscle contractile and non-contractile tissue with function, strength, and age in boys with Duchenne muscular dystrophy. Neuromuscul Disord. 2012 Jan;22(1):16-25. doi: 10.1016/j.nmd.2011.06.750. Epub 2011 Jul 31. PMID 21807516
- [Background] Forbes SC, Walter GA, Rooney WD, Wang DJ, DeVos S, Pollaro J, Triplett W, Lott DJ, Willcocks RJ, Senesac C, Daniels MJ, Byrne BJ, Russman B, Finkel RS, Meyer JS, Sweeney HL, Vandenborne K. Skeletal muscles of ambulant children with Duchenne muscular dystrophy: validation of multicenter study of evaluation with MR imaging and MR spectroscopy. Radiology. 2013 Oct;269(1):198-207. doi: 10.1148/radiol.13121948. Epub 2013 May 21. PMID 23696684
- [Background] Triplett WT, Baligand C, Forbes SC, Willcocks RJ, Lott DJ, DeVos S, Pollaro J, Rooney WD, Sweeney HL, Bonnemann CG, Wang DJ, Vandenborne K, Walter GA. Chemical shift-based MRI to measure fat fractions in dystrophic skeletal muscle. Magn Reson Med. 2014 Jul;72(1):8-19. doi: 10.1002/mrm.24917. Epub 2013 Sep 4. PMID 24006208
- [Background] Willcocks RJ, Arpan IA, Forbes SC, Lott DJ, Senesac CR, Senesac E, Deol J, Triplett WT, Baligand C, Daniels MJ, Sweeney HL, Walter GA, Vandenborne K. Longitudinal measurements of MRI-T2 in boys with Duchenne muscular dystrophy: effects of age and disease progression. Neuromuscul Disord. 2014 May;24(5):393-401. doi: 10.1016/j.nmd.2013.12.012. Epub 2014 Jan 11. PMID 24491484
- [Background] Arpan I, Willcocks RJ, Forbes SC, Finkel RS, Lott DJ, Rooney WD, Triplett WT, Senesac CR, Daniels MJ, Byrne BJ, Finanger EL, Russman BS, Wang DJ, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Examination of effects of corticosteroids on skeletal muscles of boys with DMD using MRI and MRS. Neurology. 2014 Sep 9;83(11):974-80. doi: 10.1212/WNL.0000000000000775. Epub 2014 Aug 6. PMID 25098537
- [Background] Arpan I, Forbes SC, Lott DJ, Senesac CR, Daniels MJ, Triplett WT, Deol JK, Sweeney HL, Walter GA, Vandenborne K. T(2) mapping provides multiple approaches for the characterization of muscle involvement in neuromuscular diseases: a cross-sectional study of lower leg muscles in 5-15-year-old boys with Duchenne muscular dystrophy. NMR Biomed. 2013 Mar;26(3):320-8. doi: 10.1002/nbm.2851. Epub 2012 Oct 9. PMID 23044995
- [Background] Forbes SC, Willcocks RJ, Triplett WT, Rooney WD, Lott DJ, Wang DJ, Pollaro J, Senesac CR, Daniels MJ, Finkel RS, Russman BS, Byrne BJ, Finanger EL, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Magnetic resonance imaging and spectroscopy assessment of lower extremity skeletal muscles in boys with Duchenne muscular dystrophy: a multicenter cross sectional study. PLoS One. 2014 Sep 9;9(9):e106435. doi: 10.1371/journal.pone.0106435. eCollection 2014. PMID 25203313
- [Background] Bendixen RM, Lott DJ, Senesac C, Mathur S, Vandenborne K. Participation in daily life activities and its relationship to strength and functional measures in boys with Duchenne muscular dystrophy. Disabil Rehabil. 2014;36(22):1918-23. doi: 10.3109/09638288.2014.883444. Epub 2014 Feb 6. PMID 24499260
- [Background] Senesac CR, Lott DJ, Forbes SC, Mathur S, Arpan I, Senesac ES, Walter GA, Vandenborne K. Longitudinal Evaluation of Muscle Composition Using Magnetic Resonance in 4 Boys With Duchenne Muscular Dystrophy: Case Series. Phys Ther. 2015 Jul;95(7):978-88. doi: 10.2522/ptj.20140234. Epub 2015 Jan 15. PMID 25592189
- [Background] Arora H, Willcocks RJ, Lott DJ, Harrington AT, Senesac CR, Zilke KL, Daniels MJ, Xu D, Tennekoon GI, Finanger EL, Russman BS, Finkel RS, Triplett WT, Byrne BJ, Walter GA, Sweeney HL, Vandenborne K. Longitudinal timed function tests in Duchenne muscular dystrophy: ImagingDMD cohort natural history. Muscle Nerve. 2018 Nov;58(5):631-638. doi: 10.1002/mus.26161. Epub 2018 Jul 24. PMID 29742798
- [Background] Chrzanowski SM, Baligand C, Willcocks RJ, Deol J, Schmalfuss I, Lott DJ, Daniels MJ, Senesac C, Walter GA, Vandenborne K. Multi-slice MRI reveals heterogeneity in disease distribution along the length of muscle in Duchenne muscular dystrophy. Acta Myol. 2017 Sep 1;36(3):151-162. eCollection 2017 Sep. PMID 29774305
- [Background] Willcocks RJ, Forbes SC, Walter GA, Vandenborne K. Magnetic resonance imaging characteristics of injection site reactions after long-term subcutaneous delivery of drisapersen. Eur J Pediatr. 2019 May;178(5):777-778. doi: 10.1007/s00431-019-03349-0. Epub 2019 Feb 21. No abstract available. PMID 30790036
- [Background] Batra A, Vohra RS, Chrzanowski SM, Hammers DW, Lott DJ, Vandenborne K, Walter GA, Forbes SC. Effects of PDE5 inhibition on dystrophic muscle following an acute bout of downhill running and endurance training. J Appl Physiol (1985). 2019 Jun 1;126(6):1737-1745. doi: 10.1152/japplphysiol.00664.2018. Epub 2019 Apr 4. PMID 30946638
- [Background] Barnard AM, Lott DJ, Batra A, Triplett WT, Forbes SC, Riehl SL, Willcocks RJ, Smith BK, Vandenborne K, Walter GA. Imaging respiratory muscle quality and function in Duchenne muscular dystrophy. J Neurol. 2019 Nov;266(11):2752-2763. doi: 10.1007/s00415-019-09481-z. Epub 2019 Jul 26. PMID 31350642
- [Background] Barnard AM, Riehl SL, Willcocks RJ, Walter GA, Angell AM, Vandenborne K. Characterizing Enrollment in Observational Studies of Duchenne Muscular Dystrophy by Race and Ethnicity. J Neuromuscul Dis. 2020;7(2):167-173. doi: 10.3233/JND-190447. PMID 31929119
- [Background] Barnard AM, Willcocks RJ, Triplett WT, Forbes SC, Daniels MJ, Chakraborty S, Lott DJ, Senesac CR, Finanger EL, Harrington AT, Tennekoon G, Arora H, Wang DJ, Sweeney HL, Rooney WD, Walter GA, Vandenborne K. MR biomarkers predict clinical function in Duchenne muscular dystrophy. Neurology. 2020 Mar 3;94(9):e897-e909. doi: 10.1212/WNL.0000000000009012. Epub 2020 Feb 5. PMID 32024675
- [Background] Rooney WD, Berlow YA, Triplett WT, Forbes SC, Willcocks RJ, Wang DJ, Arpan I, Arora H, Senesac C, Lott DJ, Tennekoon G, Finkel R, Russman BS, Finanger EL, Chakraborty S, O'Brien E, Moloney B, Barnard A, Sweeney HL, Daniels MJ, Walter GA, Vandenborne K. Modeling disease trajectory in Duchenne muscular dystrophy. Neurology. 2020 Apr 14;94(15):e1622-e1633. doi: 10.1212/WNL.0000000000009244. Epub 2020 Mar 17. PMID 32184340
- [Background] Forbes SC, Arora H, Willcocks RJ, Triplett WT, Rooney WD, Barnard AM, Alabasi U, Wang DJ, Lott DJ, Senesac CR, Harrington AT, Finanger EL, Tennekoon GI, Brandsema J, Daniels MJ, Sweeney HL, Walter GA, Vandenborne K. Upper and Lower Extremities in Duchenne Muscular Dystrophy Evaluated with Quantitative MRI and Proton MR Spectroscopy in a Multicenter Cohort. Radiology. 2020 Jun;295(3):616-625. doi: 10.1148/radiol.2020192210. Epub 2020 Apr 14. PMID 32286193
- [Background] Barnard AM, Willcocks RJ, Finanger EL, Daniels MJ, Triplett WT, Rooney WD, Lott DJ, Forbes SC, Wang DJ, Senesac CR, Harrington AT, Finkel RS, Russman BS, Byrne BJ, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Skeletal muscle magnetic resonance biomarkers correlate with function and sentinel events in Duchenne muscular dystrophy. PLoS One. 2018 Mar 19;13(3):e0194283. doi: 10.1371/journal.pone.0194283. eCollection 2018. PMID 29554116
- [Background] Willcocks RJ, Triplett WT, Forbes SC, Arora H, Senesac CR, Lott DJ, Nicholson TR, Rooney WD, Walter GA, Vandenborne K. Magnetic resonance imaging of the proximal upper extremity musculature in boys with Duchenne muscular dystrophy. J Neurol. 2017 Jan;264(1):64-71. doi: 10.1007/s00415-016-8311-0. Epub 2016 Oct 24. PMID 27778157
- [Background] Forbes SC, Willcocks RJ, Rooney WD, Walter GA, Vandenborne K. MRI quantifies neuromuscular disease progression. Lancet Neurol. 2016 Jan;15(1):26-8. doi: 10.1016/S1474-4422(15)00320-8. Epub 2015 Nov 6. No abstract available. PMID 26549781
- [Background] Lott DJ, Taivassalo T, Senesac CR, Willcocks RJ, Harrington AM, Zilke K, Cunkle H, Powers C, Finanger EL, Rooney WD, Tennekoon GI, Vandenborne K. Walking activity in a large cohort of boys with Duchenne muscular dystrophy. Muscle Nerve. 2021 Feb;63(2):192-198. doi: 10.1002/mus.27119. Epub 2020 Nov 27. PMID 33188573
- [Background] Senesac CR, Barnard AM, Lott DJ, Nair KS, Harrington AT, Willcocks RJ, Zilke KL, Rooney WD, Walter GA, Vandenborne K. Magnetic Resonance Imaging Studies in Duchenne Muscular Dystrophy: Linking Findings to the Physical Therapy Clinic. Phys Ther. 2020 Oct 30;100(11):2035-2048. doi: 10.1093/ptj/pzaa140. PMID 32737968
- [Background] Barnard AM, Hammers DW, Triplett WT, Kim S, Forbes SC, Willcocks RJ, Daniels MJ, Senesac CR, Lott DJ, Arpan I, Rooney WD, Wang RT, Nelson SF, Sweeney HL, Vandenborne K, Walter GA. Evaluating Genetic Modifiers of Duchenne Muscular Dystrophy Disease Progression Using Modeling and MRI. Neurology. 2022 Nov 22;99(21):e2406-e2416. doi: 10.1212/WNL.0000000000201163. Epub 2022 Sep 2. PMID 36240102
- [Background] Nair KS, Lott DJ, Forbes SC, Barnard AM, Willcocks RJ, Senesac CR, Daniels MJ, Harrington AT, Tennekoon GI, Zilke K, Finanger EL, Finkel RS, Rooney WD, Walter GA, Vandenborne K. Step Activity Monitoring in Boys with Duchenne Muscular Dystrophy and its Correlation with Magnetic Resonance Measures and Functional Performance. J Neuromuscul Dis. 2022;9(3):423-436. doi: 10.3233/JND-210746. PMID 35466946
- [Background] Finkel RS, Finanger E, Vandenborne K, Sweeney HL, Tennekoon G, Shieh PB, Willcocks R, Walter G, Rooney WD, Forbes SC, Triplett WT, Yum SW, Mancini M, MacDougall J, Fretzen A, Bista P, Nichols A, Donovan JM. Disease-modifying effects of edasalonexent, an NF-kappaB inhibitor, in young boys with Duchenne muscular dystrophy: Results of the MoveDMD phase 2 and open label extension trial. Neuromuscul Disord. 2021 May;31(5):385-396. doi: 10.1016/j.nmd.2021.02.001. Epub 2021 Feb 4. PMID 33678513
- [Background] Willcocks RJ, Forbes SC, Walter GA, Sweeney L, Rodino-Klapac LR, Mendell JR, Vandenborne K. Assessment of rAAVrh.74.MHCK7.micro-dystrophin Gene Therapy Using Magnetic Resonance Imaging in Children With Duchenne Muscular Dystrophy. JAMA Netw Open. 2021 Jan 4;4(1):e2031851. doi: 10.1001/jamanetworkopen.2020.31851. PMID 33394000
- [Background] Barnard AM, Lott DJ, Batra A, Triplett WT, Willcocks RJ, Forbes SC, Rooney WD, Daniels MJ, Smith BK, Vandenborne K, Walter GA. Characterizing Expiratory Respiratory Muscle Degeneration in Duchenne Muscular Dystrophy Using MRI. Chest. 2022 Mar;161(3):753-763. doi: 10.1016/j.chest.2021.08.078. Epub 2021 Sep 15. PMID 34536384
- [Background] Willcocks RJ, Barnard AM, Wortman RJ, Senesac CR, Lott DJ, Harrington AT, Zilke KL, Forbes SC, Rooney WD, Wang DJ, Finanger EL, Tennekoon GI, Daniels MJ, Triplett WT, Walter GA, Vandenborne K. Development of Contractures in DMD in Relation to MRI-Determined Muscle Quality and Ambulatory Function. J Neuromuscul Dis. 2022;9(2):289-302. doi: 10.3233/JND-210731. PMID 35124659
- [Background] Mercuri E, Vilchez JJ, Boespflug-Tanguy O, Zaidman CM, Mah JK, Goemans N, Muller-Felber W, Niks EH, Schara-Schmidt U, Bertini E, Comi GP, Mathews KD, Servais L, Vandenborne K, Johannsen J, Messina S, Spinty S, McAdam L, Selby K, Byrne B, Laverty CG, Carroll K, Zardi G, Cazzaniga S, Coceani N, Bettica P, McDonald CM; EPIDYS Study Group. Safety and efficacy of givinostat in boys with Duchenne muscular dystrophy (EPIDYS): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2024 Apr;23(4):393-403. doi: 10.1016/S1474-4422(24)00036-X. PMID 38508835
- [Background] Willcocks RJ, Barnard AM, Daniels MJ, Forbes SC, Triplett WT, Brandsema JF, Finanger EL, Rooney WD, Kim S, Wang DJ, Lott DJ, Senesac CR, Walter GA, Sweeney HL, Vandenborne K. Clinical importance of changes in magnetic resonance biomarkers for Duchenne muscular dystrophy. Ann Clin Transl Neurol. 2024 Jan;11(1):67-78. doi: 10.1002/acn3.51933. Epub 2023 Nov 6. PMID 37932907
- [Background] Kim S, Willcocks RJ, Daniels MJ, Morales JF, Yoon DY, Triplett WT, Barnard AM, Conrado DJ, Aggarwal V, Belfiore-Oshan R, Martinez TN, Walter GA, Rooney WD, Vandenborne K. Multivariate modeling of magnetic resonance biomarkers and clinical outcome measures for Duchenne muscular dystrophy clinical trials. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1437-1449. doi: 10.1002/psp4.13021. Epub 2023 Aug 27. PMID 37534782
- [Background] Yoon DY, Daniels MJ, Willcocks RJ, Triplett WT, Morales JF, Walter GA, Rooney WD, Vandenborne K, Kim S; DMD MR Biomarker Steering Committee. Five multivariate Duchenne muscular dystrophy progression models bridging six-minute walk distance and MRI relaxometry of leg muscles. J Pharmacokinet Pharmacodyn. 2024 Dec;51(6):671-683. doi: 10.1007/s10928-024-09910-1. Epub 2024 Apr 12. PMID 38609673
- See also: active website — http://www.imagingNMD.org